CLINICAL TRIAL: NCT03837886
Title: Sodium Bicarbonate Supplementation Promotes Changes in Performance, Muscle Activity and Strength of Individuals Trained During the Performance of Intermittent and Intense Task? Randomized, Double-blind, Crossover Trial
Brief Title: Effects of Sodium Bicarbonate Supplementation on Intermittent and Intense Task
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Collaborators: Marcelo Martins Kalytczak (Unknown)
Responsible Party: Principal Investigator, Fabiano Politti, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: FP001
Record Dates: First submitted 2019-02-06; First posted 2019-02-12 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Sodium Bicarbonate; Alkalosis, Metabolic; Electromyography; Fatigue
MeSH Terms: conditions — Alkalosis; Fatigue | interventions — Sodium Bicarbonate; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alkalosis group (Experimental): The subjects should receive gelatinous capsules containing 0.3 g.kg -1 of sodium bicarbonate
  Interventions: Dietary Supplement: Sodium bicarbonate
- Placebo group (Placebo Comparator): The subjects should receive gelatinous capsules containing 0.3 g.kg -1 of Calcium Carbonate
  Interventions: Dietary Supplement: Calcium carbonate

INTERVENTIONS:
Dietary Supplement: Sodium bicarbonate — The subjects should ingest 0.3g.kg of sodium bicarbonate 90 minutes before the beginning of the protocol task.
  Arms: Alkalosis group
Dietary Supplement: Calcium carbonate — The subjects should receive gelatinous capsules containing 0.3 g.kg -1 of Calcium Carbonate
  Arms: Placebo group

SUMMARY:
The aim of this study was to verify if sodium bicarbonate (NaHCO3) suplementation promotes changes in the performance, muscular activity and strength of individuals trained during the intermittent and intense task . Twelve trained adult men will participate in this randomized, double-blind, crossover clinical trial. Each participant should receive two types of intervention with a 14-day interval between conditions: alkalosis (ALK) in which gelatinous capsules containing 0.3 g.kg -1 of NaHCO 3 and placebo (PLA) are administered, in which 0.3 g.kg-1 of Calcium Carbonate (CaCO3). The following results will be considered: electromyographic activity (EMG) of the quadriceps muscle, peak torque, pH, lactate, and perception of effort, recovery and pain questionnaires, which will be collected during intermittent and high intensity DI protocol. ANOVA of repeated measures will be used to verify possible differences between groups.

ELIGIBILITY:
Inclusion Criteria:

* resistance trained men (minimum 12 moths resistance training experience)

Exclusion Criteria:

* diabetes mellitus;
* respiratory (asthma, COPD), renal, metabolic, rheumatic and cardiovascular disorders;
* acid-base balance disorder;
* continuous use of some type of medication;
* use of high-protein supplementation and creatine supplementation;
* users of anabolic steroids.

Ages: 20 Years to 42 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-10-20 (Estimated); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Electromyographic activity of the femoral quadriceps evaluated with electromyography equipment | 60 minutes
  The electromyographic activity will be obtained during the execution of 10 series composed of ten repetitions of extension (concentric phase) and flexion (eccentric phase) of the knee joint, at an angular velocity of 120os-1 (radians per second), with interval of 1 minute interval between sets in an isokinetic dynamometer.
Peak torque assessed with isokinetic dynamometer equipment | 60 minutes
  The peak torque will be obtained during the execution of 10 series composed of ten repetitions of extension (concentric phase) and flexion (eccentric phase) of the knee joint, at an angular velocity of 120os-1 (radians per second), with interval of 1 minute interval between sets.

SECONDARY OUTCOMES:
Lactate assessed with portable lactometer | 15 seconds
  The lactate quantification will be performed before and after the test session characterized by the execution of 10 series composed of ten repetitions of extension (concentric phase) and flexion (eccentric phase) of the knee joint, at an angular velocity of 120os-1 (radians per second), with an interval of 1 minute between sets in an isokinetic dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Nove de Julho University, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided